CLINICAL TRIAL: NCT02546206
Title: Influence of Probiotics on Clinical Parameters and GCF Levels of Interleukin-1β in Experimental Gingivitis: a Randomized Controlled Clinical Trial
Brief Title: Probiotic Yoghurt Effect on Experimental Gingivitis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MAR-2011-10-11/14
Record Dates: First submitted 2015-08-30; First posted 2015-09-10 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-08

CONDITIONS: Gingivitis
Keywords: Bifidobacterium; Gingivitis; Gingival crevicular fluid; Interleukin-1beta; Probiotics
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic Yoghurt (Experimental): Probiotic yoghurt consumption
  Interventions: Dietary Supplement: Probiotic Yoghurt
- Natural Yoghurt (Placebo Comparator): Natural yoghurt consumption
  Interventions: Dietary Supplement: Natural Yoghurt

INTERVENTIONS:
Dietary Supplement: Probiotic Yoghurt — Probiotic yoghurt consumption
  Arms: Probiotic Yoghurt
Dietary Supplement: Natural Yoghurt — Natural yoghurt consumption
  Arms: Natural Yoghurt

SUMMARY:
The aim of this study was to evaluate the effects of probiotic yoghurt on the development of gingival inflammation.

Fifty-one periodontally healthy individuals were given standard oral hygiene instructions and randomly divided into two groups. The test group subjects (n=26) consumed probiotic yoghurt containing Bifidobacterium animalis subsp. lactis and the control subjects (n=25) natural yoghurt for 28 days. Following yoghurt consumption, mechanical plaque control was interrupted for the next 5 days in both groups. Gingival crevicular fluid (GCF) samples and clinical data (consisted of plaque and gingival indices, probing depth, bleeding on probing) were collected at baseline, after 28 and 33 days. Interleukin-1β levels were determined in GCF by ELISA.

DETAILED DESCRIPTION:
Probiotics are viable bacteria with scientifically confirmed health benefits for gastrointestinal system. However, there is paucity of information on its impact in periodontal disease. The aim of this study was to evaluate the effects of probiotic yoghurt on the development of gingival inflammation.

Fifty-one periodontally healthy individuals were given standard oral hygiene instructions and randomly divided into two groups. The test group subjects (n=26) consumed probiotic yoghurt containing Bifidobacterium animalis subsp. lactis and the control subjects (n=25) natural yoghurt for 28 days. Following yoghurt consumption, mechanical plaque control was interrupted for the next 5 days in both groups. Gingival crevicular fluid (GCF) samples and clinical data (consisted of plaque and gingival indices, probing depth, bleeding on probing) were collected at baseline, after 28 and 33 days. Interleukin-1β levels were determined in GCF by ELISA.

ELIGIBILITY:
Inclusion Criteria:

* No or minimal clinical signs of gingival inflammation
* Gingival Index ≤ 1
* No probing depth (Probing depth > 3 mm)
* No approximal attachment loss > 2 mm
* Non smokers

Exclusion Criteria:

* Systemic diseases
* Antibiotics and anti-inflammatory drugs within 3 months before the study
* Untreated caries lesions or local retention factors
* Mouth-breathing
* Allergies
* Previous probiotic supplements in diet

Ages: 16 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 51 (Actual)
Dates: Start 2011-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Bleeding on probing | 33 days after yoghurt consumption
  Bleeding on probing is defined as presence of bleeding from gingival sulcus during the probing of this area via periodontal probe.

SECONDARY OUTCOMES:
Gingival Index | 33 days after yoghurt consumption
  Each of the buccal, mesial, lingual and distal surfaces of the gingival tissues is given a score of 0-3. (0 = Normal gingiva. 1 = Mild inflammation - slight change in color, slight edema. No bleeding on probing. 2. Moderate inflammation - redness, edema and glazing. Bleeding on probing. 3. Severe inflammation -marked redness and edema.)
Plaque Index | 33 days after yoghurt consumption
  Each of the four surfaces of the teeth (buccal, lingual, mesial and distal) is given a score from 0-3. (0 = No plaque in the gingival area. 1 = A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may only be recognized by running a probe across the tooth surface. 2 = Moderate accumulation of soft deposits within the gingival pocket, on the gingival margin and/or adjacent tooth surface, which can be seen by the naked eye. 3 = Abundance of soft matter within the gingival pocket and/or on the gingival margin and adjacent tooth surface. Tendency to spontaneous bleeding.)

OTHER OUTCOMES:
Probing Depth | 33 days after yoghurt consumption
  Probing depth is defined as the distance from the free gingival margin to the bottom of the periodontal pocket.
Gingival crevicular fluid Interleukin-1beta levels | 33 days after yoghurt consumption

CONTACTS AND LOCATIONS:
Overall Officials: Tuğçe Yalnızoğlu, PhD, Principal Investigator — Marmara University, Faculty of Dentistry, Department of Periodontology; Bahar Kuru, Prof Dr, Study Director — Marmara University, Faculty of Dentistry, Department of Periodontology
Locations (1):
- Marmara University, Faculty of Dentistry, Department of Periodontology, Istanbul, Sisli/Nisantasi, Turkey (Türkiye)